CLINICAL TRIAL: NCT02349256
Title: Somatoform Disorder in British South Asians - What Are the Patients' Views?
Brief Title: Somatoform Disorder in British South Asians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Global Health Primary Care Research and Innovation and Network (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: 123389
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Somatic Syndrome Disorder
Keywords: MUS; British South Asians; Somatic Symptoms; Qualitative interviews
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosed with Somatic Syndrome Disorder: Group of participants that are screened and meet criteria for diagnosis of Somatic Syndrome disorder will be asked if they wish to take part in a 1-1 qualitative interview with the researcher.

SUMMARY:
The study uses in depth interviews to understand their experience of somatoform disorder, possible explanations and their experience of somatoform disorder, possible explanations and their understanding of treatments, especially their ideas about psychosocial treatments.

DETAILED DESCRIPTION:
"Somatoform" or "functional" syndromes are those that present with physical symptoms, not explained by well-recognized medical illness. Such symptoms are common in all settings and studies have reported that they accounted for one-fifth of all new presentations in primary care. Literature suggests that they are associated with significant levels of psychological distress, disability, impairments in quality of life and high levels of healthcare utilization. Research also suggests that medically unexplained symptoms cause similar (or higher) levels of disability than medically explained symptoms in primary care settings. There have been a number of studies that have looked at the cognitive and behavioural basis of somatisation, and treatment strategies have been trialed based upon a cognitive behavior therapy (CBT)-led approach for these patients.

In British South Asian patients the difficulties in managing this condition are further compounded as culture can have an important role in shaping the experience, interpretation & clinical presentation of emotional distress. Patel reported that GPs found it very challenging to manage South Asian patients with chronic pain due to the way they present with pain, and a greater likelihood of psychosomatic presentations. Language differences as well as cultural differences contributed to the challenges, especially among first- generation South Asians. Further, they felt that self-management strategies were difficult to address. The author concludes by saying 'cultural influences play an important role in the consultation process where patients' behaviour is often bound in their cultural view of health care. (South Asian) patients' presentation of their condition makes diagnosis difficult but can also lead to miscommunication'.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of self-ascribed British South Asian origin.
* Over the age of 18 years.
* Able to understand spoken and written English and/or Urdu, Gujarati.
* Able to provide written informed consent.
* Registered with the GP practice.
* criteria for somatoform disorder (determined by PHQ15).

Exclusion Criteria:

* individuals with diagnosed physical or learning disability
* any form of psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women self ascribed British South Asian Origin .
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview | 1
  Individual qualitative interviews with a group of British South Asians to explore their understanding of somatoform disorder and available therapies. These findings will then be used to inform the development of culturally adapted Cognitive Behaviour Therapy (CBT) for somatisation in British South Asians.

CONTACTS AND LOCATIONS:
Overall Officials: Saif Bhojani, Study Chair — Research Manager
Locations (1):
- Shifa Surgery, Blackburn, United Kingdom